CLINICAL TRIAL: NCT04695366
Title: The Potential of Patient-reported Outcome Measures in Detection of Relapse in Diffuse Large B-cell Lymphoma - a Prospective Cohort Study
Brief Title: The Potential of Patient-reported Outcome Measures in Detection of Relapse in Diffuse Large B-cell Lymphoma
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Lars Møller Pedersen, Chief Physician, Head of research, PhD, MD, Herlev Hospital
Other Study IDs: LyPRO1
Record Dates: First submitted 2020-12-15; First posted 2021-01-05 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Diffuse Large B Cell Lymphoma; Patient Reported Outcome
Keywords: follow-up; surveillance; feasibility
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diffuse large B-cell lymphoma patients in year 1 and 2 of clinical follow-up: Patients (Diffuse Large B-cell Lymphoma) in complete remission after primary treatment and entering the regular follow-up program at the clinic. Baseline is defined as date of end-of-treatment visit.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Annually some 450 patients are diagnosed with Diffuse Large B-cell Lymphoma (DLBCL), in Denmark. The majority of these patients are cured with immunochemotherapy, but up to 30 % will relapse, pointing to the need for targeted surveillance and follow-up strategy. However, this strategy is constantly under debate illustrated by the missing data supporting scheduled face-to-face meetings with a clinician and routine surveillance scans in order to detect relapse. On top of the clinical problems comes the psychological burden for patients enrolled in routine surveillance. This points to the need for the development of evidence-based follow-up programs both in terms of content, regularity and assignment of responsibility between the health system and the patient. In a prospective cohort study, the investigators will collect Patient Reported Outcome (PRO) measures investigating if questionnaires can be used to detect relapse in DLBCL patients. Furthermore psychological aspects of follow-up are explored.

DETAILED DESCRIPTION:
In the Western world, DLBCL is the most common subtype of non-Hodgkin lymphoma (NHL). In Denmark, approximately 450 patients are diagnosed with DLBCL every year. Treatment with anthracycline-based immunochemotherapy (most commonly rituximab, cyclophosphamide, doxorubicin, vincristine and prednisone) is curative in the majority of DLBCL patients but a significant number of patients (up to 30 %) do not achieve a complete response (CR), and an additional subset of patients ultimately relapse after CR.

Second-line treatment with salvage chemotherapy followed by autologous hematopoietic cell transplantation (auto-HCT) is potentially curative, therefore surveillance for relapse is important.

Risk of relapse is declining after two years and for patients achieving event-free survival for 24 months (post treatment), survival beyond this timepoint is close to equivalent to that of the general population.

However optimal means of follow-up for patients with DLBCL remain controversial and have been a somewhat overlooked and contentious issue.

Traditionally, routine follow-up in DLBCL patients consists of face-to-face meetings with a specialist in an outpatient clinic, with varying intervals and a mixture of surveillance components, such as clinical examinations, blood tests or imaging procedures.

To illustrate the lack of consistency in this patient group, the ESMO guidelines recommend follow-up with 4 visits in the first year, every 6 months the next 2 years and then annually, whereas The British Society of Hematology guidelines recommend clinical follow-up for 2 years followed by discharge. Guidelines from the Danish Lymphoma Group (DLG) reflect the recommendations outlined in the Lugano classification. Patients with International Prognostic Index (IPI) 0-1 who have obtained complete remission (CR), are recommended to be followed every 3 to 4 months the first year, then every 6 months for 2 years, without routine use of image diagnostics. For patients with IPI> = 2, clinical follow-up is recommended every 3 to 4 months the first 2 years, then every 6 months for 3 years. CT scan is used 6, 12 and 24 months after completion of treatment.

In recent years the value of post-therapy surveillance scans in DLBCL has been questioned. Only a minority of relapses are detected solely via imaging and no survival advantage associated with the use of surveillance imaging has been demonstrated.

Another argument against scheduled follow-up is, that the majority of relapses are probably identified outside the scheduled follow-up visits, and by patients themselves rather than by the physicians.

Patient-reported outcome (PRO) data is information reported through questionnaires, directly by patients, about how they observe symptoms, physical function and quality of life. During recent years, PRO has experienced much attention due to the increasing evidence of the positive effect of clinical responses to PRO measures, that are applied as intervention aids both in terms of relieving the symptom burden, improvements in the overall psychosocial function of the patient and survival benefits in two studies. It has been argued that the use of PRO offers an opportunity to facilitate a transition to a more patient centred approach by strengthening the role of patients in observing themselves. But there are several barriers for the implementation of PRO, such as accessibility, user-friendliness, processing the collected information, difficulties for patients having few resources and finally the interpretation of the PRO data.

To the investigator's knowledge, no study has investigated, if collection of PRO data is useful in detection of relapse in DLBCL or other lymphoma subtypes. As of today, most studies in this patient group have focused on HRQOL, late-effects or unmet needs in survivorship after treatment of lymphoma.

To solve this dilemma between ineffective, scheduled follow-up visits and the constant need for identifying patients at risk of relapse, it has been suggested, that PRO measures offer a potential for use by clinicians as a decision aid in identifying patients in need for clinical consultation.

Psychosocial distress (anxiety, fear and depressive feelings) have been described to be significant in lymphoma survivors and associated to a more frequent use of Health Care services. One explanation is that lymphoma survivors need for psychosocial support is not met in the current follow-up program.

Another explanation, is that there may be a psychological burden to routine surveillance and scheduled follow-up visits in the outpatient clinic. Anxiety symptoms, depressive feelings and fear of recurrence (FCR) in long-term lymphoma survivors are especially prevalent in the time leading up to surveillance scans.

A fear of relapse might be a rational response after treatment of a life-threatening disease, but FCR have been associated to lower quality of life, increased psychological distress, dissatisfaction with care, and severe FCR even with an inferior overall survival compared with survivors without severe FCR.

Interestingly, it has been argued whether FCR is a consequence or a cause of anxiety, depression and lower quality of life. Maybe cancer survivors with certain anxiety traits and/or a tendency of negative views about their health and quality of life are more at risk of experiencing FCR during their survivorship.

Socio-demographic data such as female gender, younger age, living alone or poor social support have been associated with increased risk of FCR, but also poorer health conditions and advanced cancer stage (26).

To the investigator's knowledge, no study has investigated the association between socio-demographic data, comorbidities, health literacy and psychosocial distress during follow-up of lymphoma patients. It offers the potential to identify patients in need of more or less support during follow-up and to move in the direction of a more personalized care of lymphoma patients.

The aim of the study is to create a PRO questionnaire and test feasibility and the potential to detect relapse in DLBCL patients.

In addition, PRO data is collected on patient experiences during follow-up and psychological aspect of survivorship.

The investigator's hope for the future is to move towards a more patient centred and individualized follow-up after treatment of lymphoma patients.

ELIGIBILITY:
Inclusion Criteria:

1. DLBCL diagnosed according to the WHO classification
2. Age >18 years at diagnosis
3. Completed curative intent first line treatment with anthracycline-containing immuno-chemotherapy with or without consolidating radiotherapy and achieved CR on end-of-treatment CT/PET-CT scan, as recorded in the medical record by the treating physician.
4. Participated in less than 2 years of follow-up without biopsy-verified relapse
5. Access to electronic communication with health authorities (e-Boks - an electronic, closed two factor authentication)
6. Able to receive an email and complete a questionnaire in Danish

Exclusion Criteria:

1. Verified lymphoma in the central nervous system (CNS)
2. Initial treatment not completed
3. CR not reached after initial treatment
4. Palliative treatment including attenuated chemotherapy
5. Undergoing anti-lymphoma treatment or treatment for other cancer.
6. Inability to read Danish or no access to electronic communication

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: From 1 January 2021 to 31 December 2022, we will invite all DLBCL patients in remission after first-line curative treatment provided at the hematology departments of Herlev hospital, Universtity of Copenhagen, and Rigshospitalet, University of Copenhagen, to participate.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Correlation between each item in the questionnaire or groups of items and subsequent relapse | 2 years
  indicators of relapse.

SECONDARY OUTCOMES:
Impact of routine follow-up on psychological distress | 2 years
  Changes in fear of recurrence questionnaire (FCRI-SF) and quality of life questionnaires (EORTC-QLQ-C30) around time of routine follow-up visit
Impact of personality on psychological distress | 2 years
  Correlation between level of uncertainty intolerance (IUS questionnaire) and quality of life (EORTC-QLQ-C30) and fear of recurrence (FCRI-SF) and correlation between health literacy (44- item questionnaire) and quality of life (EORTC-QLQ-C30) and fear of recurrence (FCRI-SF).
Feasibility testing of electronic use of questionnaires in DLBCL patients | 2 years
  Patient compliance measured as patient satisfaction from a questionnaire and inclusion rate

CONTACTS AND LOCATIONS:
Overall Officials: Therese Lassen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Therese Lassen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No